CLINICAL TRIAL: NCT05519384
Title: Safety and Preliminary Efficacy of JK500 Cell Injection in Relapsed/Refractory Pediatric Acute Myeloid Leukemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Bejing Institute for Stem Cell and Regenerative Medicine (Unknown); Institute for Stem cell and Regeneration, Chinese Academy of Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISCRNK01001
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia, Childhood; Relapsed Leukemia; Refractory Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Intervention Model Description: They were divided into three dose groups: 10^6, 5x10^6 and 3x10^7 JK500 cells injection /kg/ time, three times a week, a total of 6 times.
  According to the principle of dose escalation, 3 patients were assigned to each dose group. After completing the treatment of 3 patients in each dose group, the Safety Review Committee (SRC) discussed whether to enter the next dose group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JK500 cell injection (Experimental): They were divided into three dose groups: 10^6, 5x10^6 and 3x10^7 JK500 cells injection /kg/ time, three times a week, a total of 6 times.
  According to the principle of dose escalation, 3 patients were assigned to each dose group. After completing the treatment of 3 patients in each dose group, the Safety Review Committee (SRC) discussed whether to enter the next dose group.
  Interventions: Drug: JK500 cell injection，cyclophosphamide，Fludarabine

INTERVENTIONS:
Drug: JK500 cell injection，cyclophosphamide，Fludarabine — After enrollment, patients received JK500 cell injection infusion after reinduction therapy. Pretreatment regimen before cell infusion: intravenous infusion of cyclophosphamide 60mg/kg day -7, intravenous infusion of fludarabine 25mg/㎡/day day -6 to -2 days. In order to activate and expand circulating NK cells, on the day of each infusion of JK500 cells, the patients were first subcutaneously injected with 100WU/ m2 of interleukin (IL)-2 0.5h-1h in advance, for a total of 6 doses.

SUMMARY:
This study is a prospective, single-center, single-arm exploratory clinical study, aiming to complete the preliminary clinical observation of 12 children with relapsed/refractory acute myeloid leukemia treated with JK500 cell injection to evaluate the safety of clinical infusion and the initial efficacy of JK500 cell injection in the treatment of children with relapsed/refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
The Main components of JK500 cell injection are regenerative natural killer (NK) cells derived from human embryonic stem cells and 0.9% sodium chloride solution.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤18, male or female;
2. Patients diagnosed as acute myeloid leukemia (AML) according to the revised World Health Organization (WHO) criteria in 2016;
3. Patients who failed to achieve CR after two standard-dose induction therapy or had recurrence within six months after CR;
4. The subject or the guardian of the subject must fully understand the purpose, nature, method and possible adverse reactions of the test, agree the subject as the subject, and sign the informed consent.

Exclusion Criteria:

1. Acute promyelocytic leukemia, chronic myelocytic leukemia, acute mixed-cell leukemia or known central nervous system leukemia;
2. AML associated with congenital syndromes such as Down syndrome, Fanconi's anemia, Bloom's syndrome, Koch's syndrome, or congenital aplastic anemia;
3. The subjects have active virus infection, and during the screening period, the serum virology test is performed, and the human immunodeficiency virus (HIV) antibody is positive, hepatitis B surface antigen or E antigen is positive, hepatitis C antibody is positive, or treponema pallidum antibody is positive;
4. Presence of active systemic infection; Participated in a drug trial within the past 4 weeks;
5. Patients who suffered from a clinically significant disease within 28 days before receiving the study product or underwent a major surgical operation within 28 days before receiving the study product, or are expected to need major surgery during the trial;
6. children with liver and kidney dysfunction, including:

   1. Serum creatinine >2× upper limit of normal reference value;
   2. Serum total bilirubin > 2× upper limit of normal reference value;
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2× upper limit of normal reference values
7. Children who have used live attenuated vaccine 4 weeks before administration or plan to use live attenuated vaccine within 6 months after administration;
8. Have any other conditions that may cause the subject to be unable to complete the study or present a significant risk to the subject in the opinion of the Investigator.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days
  DLT evaluation is defined as adverse events or laboratory abnormalities that occur within 4 weeks after investigational drug administration, are unrelated to external causes such as progressive disease, concomitant disease, and concomitant medications, including hematologic and non-hematologic adverse events (grade according to NCI CTCAE 5.0).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  ORR was defined as complete response (CR)+ incomplete bone marrow recovery (CRi) + partial response (PR). Treatment response will be assessed periodically until the end of treatment and up to 24 months after the first injection.
Minimal Residual Disease (MRD) | 24 months
  To observe the MRD status in bone marrow.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, CAMS & PUMC
Locations (1):
- Department of Pediatrics, Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No